CLINICAL TRIAL: NCT00456456
Title: The Daily Habits Survey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: American University (Other)
Other Study IDs: Study 013
Record Dates: First submitted 2007-04-03; First posted 2007-04-05 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2007-04

CONDITIONS: Food Consumption, Sleep, and Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Online survey for 11-17 year olds about behavior, sleep, and food consumption patterns. This survey can be completed on any computer that has internet access.

DETAILED DESCRIPTION:
The following opportunity is a reserach project at the American University Behavioral Pharmacology and Health Promotions Laboratory (BPHP). The study population is 11-17 year olds. The 30 minute online survey asks questions about behavior, sleep, and typical food consumption. The purpose of this survey is to better understand these habits in young people and the effects of these habits on behavior and sleep. This information will provide us with a better understanding of the daily habits in young people and guide the direction of future research projects.

ELIGIBILITY:
Inclusion Criteria:

* 11-17 years old

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300
Dates: Start 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Britta Anderson, BA, Principal Investigator — American University; Laura Juliano, PhD, Study Chair — American University
Locations (1):
- American University, Washington D.C., District of Columbia, United States